CLINICAL TRIAL: NCT03799094
Title: Clinical Outcomes of Intravenous Vitamin C Synergy With Tyrosine Kinase Inhibitor in Lung Adenocarcinoma Patients With Epidermal Growth Factor Receptor Mutations
Brief Title: Vitamin C and Tyrosine Kinase Inhibitor in Lung Cancer Patients With Epidermal Growth Factor Receptor Mutations
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clifford Hospital, Guangzhou, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2/2018-19
Record Dates: First submitted 2019-01-02; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: tyrosine kinase inhibitor; Vitamin C; non-small cell lung cancer; progression-free survival; overall survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ascorbic Acid; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 75 patients received a weekly intravenous Vitamin C injection (dose: 30 g / time, once a week, treatment termination when the disease progress is confirmed) in combination with daily taking tyrosine kinase inhibitor.
  Interventions: Drug: Vitamin C; Drug: Tyrosine kinase inhibitor
- Control group (Experimental): 75 patients received tyrosine kinase inhibitor daily. (dose: Osimertinib 80 mg/d, or Tarceva 150 mg/d, or Iressa 0.25 g/d.)
  Interventions: Drug: Tyrosine kinase inhibitor

INTERVENTIONS:
Drug: Vitamin C — Participants will receive intravenous vitamin C therapy at the indicated dose.
  Other Names: Sodium Ascorbate
  Arms: Experimental group
Drug: Tyrosine kinase inhibitor — Participants will receive Tyrosine kinase inhibitor therapy in cycles: continuous treatment at the indicated dose.

SUMMARY:
This trial was to explore whether intravenous vitamin C can prolong resistance time of Tyrosine Kinase Inhibitor(TKI) on lung adenocarcinoma patients with Epidermal Growth Factor Receptor(EGFR) mutations, and can benefit NSCLC patients.

DETAILED DESCRIPTION:
The effects of vitamin C in combination with tyrosine kinase inhibitor on tumor size, tumor markers, inflammatory factor levels, quality of life, duration of resistance, progression-free survival, and overall survival time were evaluated.

This trial is a low risk treatment, and has developed the appropriate safety measures and contingency plans to ensure patients' safety in the whole process.

Patients will be followed up after the end of the trial, and follow-up observations will be performed every month during the first year. Followed every 3 months in the second year for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Primary non-small cell lung cancer (adenocarcinoma) with EGFR mutations on exons 19 and 21.
* 18 years old to 75 years old.
* During the trial, patients were prescribed TKI drugs(received initial treatment within 2 months, or change medication within 2 months) and did not receive chemotherapy or radiotherapy at the same time.
* Eastern Cooperative Oncology Group (ECOG) performance status are 0 to 2.
* Expected survival over 3 months.
* Household registration is Guangdong Province.

Exclusion Criteria:

* Co-morbid conditions that affect survival: end stage congestive heart failure, unstable angina, myocardial infarction (within the past 6 weeks), and uncontrolled blood sugars of greater than 300 mg/dL, known chronic active hepatitis or cirrhosis.
* Glucose-6-phosphate dehydrogenase deficiency (G6PD) (a relative contraindication).
* Patients who are allergic to vitamin C.
* Patients with HIV and other infectious diseases.
* Patients who are taking anticoagulants and have coagulopathy;
* Combine dysfunction of important organs such as heart, lung, liver and kidney;
* Patients with impaired renal function (serum creatinine content > 1.2 mg/dL)
* Compromised liver function with evidence of Serum total bilirubin content, Serum alanine aminotransferase(ALT) and aspartate transaminase(AST)> 2 times normal reference value.
* Pregnant or lactating female.
* Smoking and alcohol abuse patients;
* Anti-infective treatment is required for systemic or localized serious infections;
* Patients with hyperuricacidemia (normal: 91-456 μmol / 24h (8-40mg / 24h));
* Wilson's disease.
* Evidence of significant psychiatric disorder by history or examination that would prevent completion of the study or preclude informed consent.
* Any condition that impairs the patients' ability to swallow, which impairs drug absorption or drug kinetic parameters, including any kind of gastrointestinal resection or surgery;
* History of surgery of visceral organs within 6 weeks before the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From the start date of treatment until the date of first documented progression or death, assessed up to 2 years
  From the start of treatment until the patient has tumor progression or death

SECONDARY OUTCOMES:
Overall survival | From the start date of treatment until the date of death from any cause, assessed up to 2 years.
  The length of time from the start of treatment for a disease until death

OTHER OUTCOMES:
Changes in Health Related Quality of Life: European Organisation for Research and Treatment of Cancer(EORTC) quality of life questionnaire(QLQ)-C30 | From the start date of treatment until the date of first documented progression or death, assessed up to 2 years
  Using QLQ-C30: Function subscales, (include physical, role, emotional, cognitive, social, global) (averaged, 0-100, higher value represent a better outcome); Symptoms subscales (include fatigue, nausea, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea) (averaged, 0-100, lower value represent a better outcome). Given at basal, 1, 2, 3, 6, 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Junwen Ou, PhD, Study Chair — Clifford Hospital
Locations (1):
- Clifford Hospital, Guangzhou, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT03799094/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT03799094/ICF_001.pdf